CLINICAL TRIAL: NCT06194266
Title: How to Support Women Already Followed Within the CSAPA Towards Risk Reduction and Management of Gynecological and Obstetric Issues
Brief Title: Supporting Women Towards Risk Reduction and Management of Gynecological and Obstetric Issues
Acronym: SF-CSAPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9021
Record Dates: First submitted 2023-12-18; First posted 2024-01-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Gynecologic Nursing
Keywords: Nursing; Obstetric; gynecology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The health of women who use drugs is a real public health issue where the midwife has an important role to play in the multidisciplinary support of the Center for Care, Support and Prevention in Addictology (CSAPA).

The main objective is to identify the needs and expectations of the women received in terms of reducing risks and damage at the gynecological and obstetric level.

ELIGIBILITY:
Eligibility Criteria:

* Adult women (≥ 18 years old)
* Followed at the Center for Care, Support and Prevention in Addictology (CSAPA) of the University Hospitals of Strasbourg
* Speaking and understanding French
* Agreeing to participate anonymously in this study

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: - Adult women (≥ 18 years old) followed at the Center for Care, Support and Prevention in Addictology (CSAPA) of the University Hospitals of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-09-17 (Actual)

PRIMARY OUTCOMES:
Retrospective description of the needs and expectations of women in terms of gyneco-obstetric risk reduction | Through study completion, an average of 1 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Addictologie - CHU de Strasbourg - France, Strasbourg, France